CLINICAL TRIAL: NCT07182773
Title: Pre-infusion Aerobic Cycling Exercise for CardioRespiratory Fitness in Cancer Patients
Acronym: PACE-CRC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Emer Guinan, Associate Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TRI CRF 24-02; AHP24MCG (Other Grant/Funding Number: Irish Cancer Society)
Record Dates: First submitted 2025-09-05; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: exercise; cardiorespiratory fitness; chemotherapy; exercise oncology
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of this study, blinding of the participants and the exercise professional delivering the intervention is not possible. The exercise physiologist completing baseline (T0) and post-intervention (T1) CPET assessments will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Arm (Experimental): The exercise programme will be prescribed at a moderate intensity (Target Heart rate: 60%-65% Heart Rate Reserve + resting heart rate) for 30 minutes immediately prior to infusion therapy, on their treatment days over 12- weeks. Exercise will be completed on a stationary cycle ergometer. Target heart rate will be adjusted to 50-55% Heart Rate Reserve + resting heart rate if patient is complaining of fatigue/nausea, is on beta-blockers or if haemoglobin <9g/dL. Heart rate monitoring by chest strap using the polar heart rate monitor will allow participants to self-regulate their exercise intensity. Participants should discontinue exercise and await medical review if they develop chest pain, dizziness or pre-syncope, cyanosis or pallor appearance, new musculoskeletal pain.
  Interventions: Behavioral: Exercise
- Education only (No Intervention): The control group will receive education on the physical activity recommendations during cancer treatment as per standard care

INTERVENTIONS:
Behavioral: Exercise — The exercise programme will be prescribed at a moderate intensity (Target Heart rate: 60%-65% Heart Rate Reserve + resting heart rate) for 30 minutes immediately prior to infusion therapy, on their treatment days over 12- weeks. Exercise will be completed on a stationary cycle ergometer. Target heart rate will be adjusted to 50-55% Heart Rate Reserve + resting heart rate if patient is complaining of fatigue/nausea, is on beta-blockers or if haemoglobin <9g/dL. Heart rate monitoring by chest strap using the polar heart rate monitor will allow participants to self-regulate their exercise intensity. Participants should discontinue exercise and await medical review if they develop chest pain, dizziness or pre-syncope, cyanosis or pallor appearance, new musculoskeletal pain.
  Arms: Exercise Arm

SUMMARY:
Background to this Research Patients who undergo cancer treatment involving chemotherapy or immunotherapy, can experience considerable reductions in their fitness levels. This is a concern, as exercise is a really important part of cancer care. Therefore delivering exercise programmes that support patients during their chemotherapy or immunotherapy treatment will be essential to helping people to maintain their fitness levels. Research is needed to examine the best way to introduce exercise into the patient pathway in a way that is convenient and patient-centred.

The Specific Questions Being Asked This research project aims to examine the effect of an exercise programme which involves exercising on the cancer treatment day ward with a physiotherapist while waiting for treatment infusion as a safe and effective way of supporting patients to keep fit and active during chemotherapy treatment. The trial will also investigate if it the prescribed moderate intensity exercise for 30 minutes is manageable for patients.

Trial Plan This project will be delivered as a randomised controlled trial. All participants enrolled on the trial will receive information and advice about physical activity during chemotherapy treatment from a physiotherapist with expertise in cancer care. The intervention arm will also complete an exercise session with the physiotherapist on the day of their infusion treatment over a period of 12 weeks.

The feasibility of this protocol has already been tested in 17 participants with very positive results. The information gained from this initial study will be used to deliver this trial, which will recruit 80 participants. It is hoped that the information gained from this research will provide a practical way of providing supervised exercise training for patients during chemotherapy or immunotherapy that is safe, expert-led and patient centred.

DETAILED DESCRIPTION:
Introduction

Cardiorespiratory fitness (CRF) is a critical health indicator that plays a significant role in predicting cancer risk and mortality. Notably, CRF often declines during infusion therapies such as chemotherapy and immunotherapy, and these declines may persist even after treatment completion. This reduction in CRF is concerning, as it may predispose patients to increased morbidity and mortality, especially given the cardiotoxic effects associated with some cancer treatments. Despite the importance of maintaining or improving CRF, the optimal timing and prescription for aerobic exercise in cancer care remain unclear. Current guidelines recommend that individuals with cancer aim for 150 minutes of moderate-intensity aerobic exercise weekly, or 75 minutes of vigorous-intensity exercise, along with twice-weekly resistance training. However, the prolonged periods of inactivity associated with infusion therapies, which often last several months, complicate adherence to these recommendations.

Aerobic exercise during cancer treatment has been shown to improve CRF, with systematic reviews indicating significant benefits in terms of physical function, fatigue reduction, and overall quality of life. Furthermore, exercise has been linked to improved cancer outcomes, including a reduced risk of cancer recurrence, lower cancer-specific mortality, and a decreased risk of all-cause mortality. Despite these benefits, adherence to exercise guidelines during cancer treatment remains low, with reports ranging from 8.5% to 34%. Barriers such as treatment side effects, fatigue, lack of knowledge, and time constraints often hinder patients from engaging in regular physical activity.

Recent studies suggest that supervised exercise performed immediately prior to infusion therapy may help mitigate these barriers, offering a structured and safe approach that could fit into patients' demanding treatment schedules. Additionally, there is emerging evidence that exercise performed during chemotherapy infusion could have beneficial physiological effects, such as improved tumour perfusion and enhanced drug delivery, potentially boosting the effectiveness of treatment. However, more research is needed to determine the optimal timing, duration, and intensity of exercise to achieve clinically meaningful benefits in this context.

As cancer incidence continues to rise, with approximately 44,000 new cancer cases reported annually in Ireland alone, the need for effective interventions that support patients during treatment is increasingly urgent. While exercise has demonstrated a range of physical, psychological, and immunological benefits, further investigation into the feasibility and impact of exercise during infusion therapy is essential to guide clinical practice. This protocol aims to address common barriers to exercise for cancer patients, based on recent systematic reviews and patient input, with the goal of enhancing patient care and outcomes through improved maintenance of CRF during treatment.

Aims and Objectives

The overall aim of this study is to examine the feasibility of delivering a supervised moderate intensity aerobic exercise intervention to patients with cancer directly before their infusion therapy.

The specific objectives are:

To determine the rate of recruitment of cancer patients willing to participate in the exercise programme during chemotherapy.

To examine the feasibility of intervention delivery, including exercise adherence, fidelity, and retention rates.

To examine if supervised moderate intensity aerobic exercise directly before infusion therapy increases and or maintains cardiorespiratory fitness in cancer patients to a greater extent than education alone.

To test the appropriateness of outcome assessments, data collection techniques, and suitability of proposed outcomes.

To monitor and record any adverse events to test the safety of the exercise intervention.

To gather feedback from patients regarding the acceptability of the exercise programme.

To examine the preliminary efficacy of the exercise programme on secondary endpoints such as fatigue, physical activity levels and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18.

Histological confirmed diagnosis of stage I to IIIc breast, ovarian, or colorectal cancer.

Scheduled to receive chemotherapy ± immunotherapy with curative intent over at least a 12-week period.

Medical clearance from oncologist to partake in regular exercise in accordance with ACSM preparticipation screening algorithm.

Able to use exercise bike independently.

Ability to provide written informed consent.

Exclusion Criteria:

* Advanced/metastatic disease.

Scheduled to receive concurrent chemoradiotherapy.

New pain or other pain that would preclude ability to use bike.

Inability to read and understand English.

Deemed unfit to proceed from results of CPET.

Unstable angina, arrhythmia, hypertension or decompensated heart failure.

Dementia or psychiatric illness which would preclude safe independent exercise.

Acute untreated embolus/infarct.

Dissecting aneurysm.

Acute myocarditis or pericarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment Rates | Enrolment (baseline)
  Recruitment rates will be calculated as the percentage of eligible participants who agreed to take part in the study. Recruitment rates will be calculated for each recruitment timepoint to determine which timepoint yields optimal recruitment. Reasons for declining recruitment will also be recorded.
Feasibility - Adherence Rates | Weeks 1 to 12
  Exercise adherence will be used to measure the degree to which the participants performed the exercise at the desired intensity and time. After each exercise session, participants will be asked to rate their perceived exertion that they actually achieved during the exercise session. This RPE will be compared to the moderate intensity (BORG 4-6) intensity prescribed to determine adherence to intensity. Heart rate data recorded during the exercise session will also be compared with target heart rate prescribed to assess adherence to intensity. The Adherence to exercise time will be calculated by recording the total number of minutes spent cycling in each session compared to the 30 minute cycling target.
Feasibility - Retention Rates | Post-intervention (12 weeks)
  Retention rates will be calculated as the number of participants completing the post intervention assessment. Reasons for dropout will also be recorded.
Feasibility - Satisfaction | Post intervention (12 weeks)
  Qualitative data will be used to analyse the overall delivery of the exercise programme and suitability of intervention characteristics. Qualitative data will be collected using satisfaction questionnaires.

SECONDARY OUTCOMES:
Cardiorespiratory Fitness | Baseline & 12 weeks
  CPETs will be performed on a cycle ergometer (h/p Cosmos model Cosmed E100) in the exercise physiology laboratory in the Beacon Orthopaedic Centre under the supervision of two exercise physiologists. The VO2peak test will be conducted on a cycle ergometer connected to the COSMED software. A standardised incremental ramp protocol will be used, commencing with a 2-minute phase of unloaded cycling. Followed by the ramped exercise phase with increases in workload (watts) to exhaustion in approximately 8-15 minutes for each individual. During CPET, Borg RPE scores will be recorded every 2 minutes and COSMED software captured the physiological measures from the breath-by-breath gas analyser with continuous monitoring of ventilation, carbon dioxide production, oxygen consumption and heart rate.
Body composition - Anthropometric measures | Baseline & 12 weeks
  Weight (kilogrammes (kg)) and height (centimetres (cm)) will be recorded by standard methods using a calibrated scales and stadiometer (Seca 704 S Wireless Column Scale With Integrated Measuring Rod). Body mass index (BMI) will be calculated as weight (kg) divided by height (metres (m2)).
Body Composition - Air Displacement Plethysmography (ADP) | Baseline & 12 weeks
  ADP will be used to determine body composition and will be performed using the 'Bod Pod'. Outputs from the Bod Pod provide multiple metrics of body composition. Measures recorded will include; fat mass, fat free mass, and skeletal muscle mass.
Health Related Quality of Life | Baseline & 12 weeks
  Health-related quality of life will be determined by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30 version 3.0) and its relevant subscales. The EORTC-QLQ-C30 manual advises that all of the scales and single item measures range in score from 0 to 100. A high score for the functional scales and functional single items represents a high/healthy level of functioning, whereas a high score for the symptom scales and symptom item represents a high level of symptom burden or problems.
Fatigue | Baseline & 12 weeks
  Fatigue will be measured using the Brief Fatigue Inventory (BFI). The BFI is a 9-item scale to assess the severity of fatigue and the impact of fatigue on daily functioning in the past 24 hours. BFI scoring guidance categorises fatigue as mild (1-3), moderate (4-6), or severe (7-10), based on a global score calculated as the average of the nine items, where 0 is no fatigue and 10 is the worst possible fatigue or complete interference. A score of 4 or greater indicates a need for intervention, and scores of 7-10 represent severe fatigue
Physical Activity Levels | Baseline & 12 weeks
  Participants self-reported physical activity levels will be recorded using The International Physical Activity Questionnaire - Short Form (IPAQ-SF). The IPAQ-SF is a 7 item open ended questionnaire on an individuals physical activity in the last 7 days. The IPAQ-SF scoring protocol involves calculating a total score in MET-minutes/week by combining walking, moderate, and vigorous activity durations, then categorising the score into low (< 600), moderate (600-3,000), or high (> 3,000 MET-minutes/week) levels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kearney N, Connolly D, Begic S, Mockler D, Guinan E. Feasibility metrics of exercise interventions during chemotherapy: A systematic review. Crit Rev Oncol Hematol. 2024 Mar;195:104272. doi: 10.1016/j.critrevonc.2024.104272. Epub 2024 Jan 23. PMID 38272152